CLINICAL TRIAL: NCT04595552
Title: Language Profile of Cochlear Implanted Children at Assiut University, Egypt
Brief Title: Language Development in Cochlear Implant Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdallah Metwally Abdelzaher, Principal invistegator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Language in cochlear implant
Record Dates: First submitted 2020-09-25; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Language; Development
Keywords: language; cochlear; implant
MeSH Terms: conditions — Language | interventions — Language Therapy

STUDY DESIGN:
Intervention Model Description: interventional prospective study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Children with cochlear implant were given Auditory training and language therapy
  Interventions: Other: language therapy

INTERVENTIONS:
Other: language therapy — auditory training and language therapy for 6 months up to 2 years in 2 session per week the duration of session 30 minuets

SUMMARY:
The aim of this work is to assess language development in cochlear implanted children in Assiut university hospital and to assess the impact of some related factors (age of implantation, family motivation and education, age of hearing loss and the pre-implanted language therapy or pre-implanted hearing aid wearing) on this development.

Adoption of newborn hearing screening programs across the nations has resulted in early identification and confirmation of hearing losses in youngest and vulnerable populations. Early identification often results in early intervention using hearing technology assistance via hearing aids or cochlear implants, parental education programs, and speech-language therapy The major goal of intervention is to capitalize on providing sensory, motor, and interactive exchanges at the earliest stages of communication development as a means of reducing the deleterious effects of auditory deprivation

DETAILED DESCRIPTION:
A cochlear implant is a device that stimulates the auditory nerve electrically to produce hearing percepts. It has an external component that receives incoming sound, processes it according to a predefined strategy, and transfers the signal across the skin. A small, implanted electronic device receives and decodes the transmitted signal and stimulates electrodes in the cochlea. The electrodes stimulate the auditory nerve directly, bypassing the hair cells that implement the first stage of auditory neural processing in normal ears. The extended use of multichannel cochlear implants in adults brought about the first major success, both scientific and commercial, of a neural sensory prosthesis that replaced a human sense with an electronic device Cochlear implants are now widely used in young deaf children and have shown tremendous promise in facilitating a variety of developmental outcomes. Specifically, improvements have been shown in oral language, speech perception and recognition, attention, and behavioral development.

Medical advances, as well as technological inventions such as digital hearing aids and cochlear implants, have made significant changes in the likelihood that a child with hearing loss will achieve adequate speech perception, intelligible speech and language competency, though none of these is yet guaranteed for all children . Despite these advances, it is probable that a child with hearing loss faces a significant delay in exposure to auditory stimulation, leading to delays in the normal course of oral language development through audition. Research findings suggest that children who received an implant even before 12 months had a one year expressive language delay . Others found variable degrees of delay with children who received implants before age 2 of years.Others found that lowering the age of implantation does seem to improve the prospects of normal language acquisition but the evidence does not suggest that children with cochlear implants perform like hearing peers on average .

Most children who are born profoundly deaf or who become deaf before the age of 3 years fall significantly behind their normal-hearing peers in their mastery of the surrounding oral language in its written, read, spoken, and signed forms.

One of the most important factors shown to influence the development of communication abilities in pediatric cochlear implant recipients is age at time of implantation .

Children implanted by 12 months of age demonstrate better language development compared with children who receive their cochlear implant between 13 and 24 months. This supports the provision of a cochlear implant within the first year of life to enhance the likelihood that a child with severe-to-profound hearing impairment will commence elementary school with age-appropriate language skills. The implanted prior to 3 years had significantly faster rates of language development than later-implanted children.

Two additional demographic factors that influence communication development in children with cochlear implants are communication mode and residual hearing. Children with prelingual deafness who use oral communication generally achieve significantly higher levels of speech perception, speech production, and/or language skills than their deaf peers who use total communication, that is, the combined use of signed and spoken language Speech perception performance with cochlear implants appears related to several factors. Higher speech perception appears linked to shorter periods of auditory deprivation, greater amounts of residual hearing, and younger ages of implantation Spoken language performance was related to the age the hearing loss was identified and the amount of typical hearing experience a child might have before losing their residual hearing

ELIGIBILITY:
Inclusion Criteria:

All these patients have satisfactory threshold of hearing post operatively proved by full post-operative audiological evaluation.

-

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
assessment of expressive language in cochlear implant children | pre therapy
  expressive language score in The Arabic language test scale prepared by Nahla Abd Elaziz Refaey 2004 in continuous number, higher value 100 and lower value 0, higher value is better outcome
assessment of receptive language in cochlear implant children | pre therapy
  receptive language score in The Arabic language test scale prepared by Nahla Abd Elaziz Refaey 2004 in continuous number, higher value 100 and lower value 0, higher value is better outcome
semantics score in language test in The continuous number | pre therapy
  semantics score in The Arabic language test scale prepared by Nahla Abd Elaziz Refaey 2004 in continuous number, higher value 100 and lower value 0, higher value is better outcome

SECONDARY OUTCOMES:
assessment of expressive language in cochlear implant children | An average of 1 year post therapy
  expressive language score in The Arabic language test scale prepared by Nahla Abd Elaziz Refaey in continuous number, higher value 100 and lower value 0, higher value mean better outcome
assessment of receptive language in cochlear implant children | An average of 1 year post therapy
  receptive language score in The Arabic language test scale prepared by Nahla Abd Elaziz Refaey in continuous number, higher value 100 and lower value 0, higher value mean better outcome
semantics score in language test in continuous number | An average of 1 year post therapy
  semantics score in The Arabic language test scale prepared by Nahla Abd Elaziz Refaey 2004 in continuous number, higher value 100 and lower value 0, higher value 100 and lower value 0

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah Abdelzaher, Dr, Principal Investigator — Assiut University
Locations (1):
- Medecine, Asyut, Egypt

REFERENCES:
- [Background] Levitt H, McGarr N, Geffner D. Development of language and communication skills in hearing-impaired children. Introduction. ASHA Monogr. 1987 Oct;(26):1-8. No abstract available. PMID 3509663
- [Background] Moeller MP, Osberger MJ, Eccarius M. Language and learning skills of hearing-impaired students. Receptive language skills. ASHA Monogr. 1986 Mar;(23):41-53. No abstract available. PMID 3730031
- [Background] Osberger MJ, Moeller MP, Eccarius M, Robbins AM, Johnson D. Language and learning skills of hearing-impaired students. Expressive language skills. ASHA Monogr. 1986 Mar;(23):54-65. No abstract available. PMID 3730032